CLINICAL TRIAL: NCT02208622
Title: Bioavailability of Zinc and Iron From a Whey-based Protein Supplement Consumed With a Habitual Plant-based Diet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Universidad Autonoma de Queretaro (Other); International Atomic Energy Agency (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: 13-0398
Record Dates: First submitted 2014-08-01; First posted 2014-08-05 (Estimated); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Nutritional Deficiency
Keywords: Zinc absorption; Iron Absorption; Whey Protein; Mexico; Stable isotopes
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Study 1: Whey Supplement Day 1 (Experimental): Children in this arm received the whey supplement as part if their diet on day 1.
  Interventions: Dietary Supplement: Study 1: Whey Supplement Day 1
- Study 1: Whey Supplement Day 2 (Experimental): Children in this arm received whey supplement as part of their diet on day 2.
  Interventions: Dietary Supplement: Study 1: Whey Supplement Day 2
- Study 2: Whey Supplement (Experimental): Children in this arm received a whey supplement as part of their diet.
  Interventions: Dietary Supplement: Study 2: Whey Supplement
- Study 2: Control (No Intervention): Children in this arm did not receive a whey supplement as part of their diet.

INTERVENTIONS:
Dietary Supplement: Study 1: Whey Supplement Day 1 — Whey supplement was given on day 1, control diet on day 2
  Arms: Study 1: Whey Supplement Day 1
Dietary Supplement: Study 1: Whey Supplement Day 2 — Control diet was given day 1, whey supplement was given day 2
  Arms: Study 1: Whey Supplement Day 2
Dietary Supplement: Study 2: Whey Supplement — Whey supplement was given as part of diet for both day 1 and 2 of study
  Arms: Study 2: Whey Supplement

SUMMARY:
Bioavailability of iron and zinc from habitual plant-based diets consumed by young children in Mexico is low due to the high phytate content. Whey protein has been found to increase zinc absorption, thus, providing a whey based supplement with micronutrients may be an effective strategy to increase iron and zinc bioavailability from plant-based foods and alleviate iron and zinc deficiencies. The investigators compared absorption of zinc and iron in children receiving diets with and without whey protein supplements (WPS).

DETAILED DESCRIPTION:
Study 1: Zinc absorption studies The zinc study employed a 2-day cross-over design, labeling the WPS diet with a different zinc stable isotope (67Zn) than the control diet (70Zn). All meals during the 2-day period were labeled with tracer. The dual isotope ratio technique was used with a 3rd Zn stable isotope (68Zn) given intravenously and urine enrichment of all isotopes measured on Study Days 6-9 to measure fractional absorption of Zn (FAZ). The amount of Zn absorbed for the day was determined by multiplying the Zn intake for the day (determined from lab analyses of duplicate test meals) by the FAZ. Children (n=16) were randomized as to the order in which they consume the test and control meals on Study Day 1 and 2.

Study 2: Iron absorption studies The iron study was a cross sectional study with one group receiving control meals and the second group receiving the same control meal plus WPS. Iron absorption was measured using the erythrocyte iron incorporation technique with labeling of all meals over 2 days (58Fe). This was preceded by a reference dose of Fe57 and ascorbate on the previous day. Children (n=32) were randomized to receive the control diet or intervention diet (control diet + WPS).

ELIGIBILITY:
Inclusion Criteria:

* 2-3 years of age
* Live in poor, rural communities
* Healthy
* Parents had provided informed consent

Exclusion Criteria:

* An acute or chronic illness which affects gut function, or
* They are breast feeding.

Ages: 2 Years to 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2013-08 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
Zinc Absorption | 2 days
  Absorption of zinc was compared in young children when given a habitual diet with and without a whey protein supplement. Fractional absorption of zinc for a day was measured by extrinsic labeling with stable isotopes of zinc. Fractional absorption of zinc was measured by a dual isotope tracer ratio technique. Measurement of total zinc in duplicate diets on test day will allow determination of quantity of this micronutrient absorbed (mg/d).
Iron Absorption | 2 days
  Absorption of iron was compared in young children when given a habitual diet with and without a whey protein supplement. Fractional absorption of iron for two days was measured by extrinsic labeling with stable isotopes of iron and measuring erythrocyte enrichment. Measurement of total iron in duplicate diets on test days will allow determination of quantity of this micronutrient absorbed (mg/d).

CONTACTS AND LOCATIONS:
Overall Officials: Michael Hambidge, MD, Principal Investigator — University of Colorado, Denver
Locations (2):
- University of Colorado Anschutz Medical Campus, Aurora, Colorado, United States
- Universidad Autonoma de Queretaro, Querétaro, Mexico